CLINICAL TRIAL: NCT01300871
Title: Alopecia Secondary to Endocrine Therapy in Postmenopausal Women With Breast Cancer
Status: Terminated | Type: Observational
Why Stopped: Poor patient accrual
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: Alopecia; 10-0906-CE (Other: Research Ethics Board)
Record Dates: First submitted 2011-02-18; First posted 2011-02-23 (Estimated); Last update posted 2014-09-26 (Estimated); Status verified 2011-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Postmenopausal Women on Endocrine Therapy: Postmenopausal women with Breast Cancer that undergo Endocrine Therapy.

SUMMARY:
This is a study to determine the prevalence and severity of alopecia (hair loss) experienced by postmenopausal breast cancer patients receiving endocrine therapy including Tamoxifen, Letrozole (Femara), Exemestane (Aromasin), or Anastrozole (Arimidex).

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women
* Diagnosed with hormone-receptor positive breast cancer
* Commenced adjuvant endocrine therapy ≥ 3 months ago, specifically Tamoxifen, Anastrozole, Exemestane, and/or Letrozole
* Good command of the English language
* Under the care of a medical oncologist at Princess Margaret Hospital

Exclusion Criteria:

* Previously received chemotherapy
* Recurrent and/or metastatic disease
* History of endocrine, dermatology, or immune system disorders known to alter hair growth (ie. Hypothyroidism and iron deficiency)

Min Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients that attend Medical Oncology Breast Clinics at Princess Margaret Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2011-01; Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Severity of Alopecia Tool (SALT) | 1 year
  The proportion of postmenopausal breast cancer patients on endocrine therapy who experience grade S1 to S5 alopecia as defined by the Severity of Alopecia Tool (SALT).

SECONDARY OUTCOMES:
Comparison of Tamoxifen, AI or Tamoxifen plus AI | 1 year
  Comparison of the proportion of postmenopausal breast cancer patients treated with Tamoxifen monotherapy, AI monotherapy, or a switch from Tamoxifen to AI who experience alopecia.
Severity of Alopecia Tool (SALT) | 1 year
  To identify the severity, or grade, of hair loss experienced by our target population. The severity of alopecia will be represented as a percentage, again in accordance with the SALT.

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay Carlsson, Principal Investigator — University Health Network-Princess Margaret Hospital
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada